CLINICAL TRIAL: NCT05996237
Title: Older Adults' Readiness to Stop Prescribed Medications with Guidance from Health Care Professionals
Brief Title: Older Adults' Readiness to Stop Prescribed Medications
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Steven M. Albert, Professor, University of Pittsburgh
Other Study IDs: STUDY23060137
Record Dates: First submitted 2023-08-09; First posted 2023-08-18 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Polypharmacy, Decision-making

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Registry participants: Participants in the University of Pittsburgh Claude D. Pepper Center community research registry. Potential participants will have stable regimens of 5+ prescribed medications and recent physician contact but no hospitalization in the prior 6 months.

SUMMARY:
Polypharmacy, regular use of 5+ prescribed medications, is common among older adults and potentially harmful. Patients differ in their concern about medications, comfort in raising questions about them, and trust and confidence in physician judgment. This pilot observational research will determine older adults' readiness to "deprescribe," that is, stop prescribed medications under physician guidance.

DETAILED DESCRIPTION:
The purpose of this research is to assess readiness to deprescribe, that is, to determine how willing patients are to stop prescriptions that may no longer be necessary or may no longer have a favorable benefit-risk ratio. This readiness depends on many factors, including a patient's trust in a health care provider, how proactive patients are in seeking care, and patients' comfort in changing longstanding medical regimens.

The proposed two-wave survey research will use validated instruments and recruit from an older adult research registry to determine (i) readiness to deprescribe at baseline, (ii) correlates of such readiness, and (iii) effects of intercurrent illness and changing health on readiness to deprescribe at 6 months.

Specific aims:

1. Determine readiness to deprescribe among a sample of patients with 5+ prescriptions using validated scales.
2. Determine correlates of readiness to deprescribe. Patients differing in age, gender, race, education, and comorbidity may differ in willingness to stop prescribed medications.
3. Determine the effect of intercurrent illness on readiness to deprescribe. Over 6 months, we anticipate some patients will have a new onset of illness or hospitalization, or increasing levels of disability. We would like to determine if these changes in medical status affect readiness to deprescribe.

ELIGIBILITY:
Inclusion Criteria:

1. 65 years or older
2. Medical visit within past 6 months
3. Self-report of at least 5 regular medications for at least 4 weeks

Exclusion criteria:

1. Diagnosis of dementia or score <=4 on Memory Impairment Screen
2. Hospitalization in prior 30 days with change in medications

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Participants in the University of Pittsburgh Claude D. Pepper communty research registry.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2023-09-21 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Patient Motivation to Deprescribe | Change over 6 months
  Self-report measure (Linsky 2020): range 1-5; high scores = greater readiness to deprescribe; mean (SD) in VA sample 2.99 (0.80)

SECONDARY OUTCOMES:
Self-reported stopping/changing prescription medication | 6 months
  Self-report of stopping, tapering, or altering use of any prescription, with or without physician discussion

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual-level data will be made available to investigators upon request following publication of key findings.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After 6/1/25, available for 2 years
Access Criteria: Written request to investigator